CLINICAL TRIAL: NCT04622800
Title: Investigation Of The Effect Of Proprioceptive Neuromuscular Fasilitation Tecniques On Muscle Strenght And Pectoralis Minor Muscle Tightness In Individuals With Scapular Dyskinesis
Brief Title: Investigation Of The Effect Of Proprioceptive Neuromuscular Fasilitation Tecniques in Scapular Dyskinesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HANDE GUNEY, Associate professor, Hacettepe University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PNF2020
Record Dates: First submitted 2020-10-30; First posted 2020-11-10 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Scapular Dyskinesis
Keywords: Scapular Dyskinesis
MeSH Terms: interventions — Exercise; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals applied with proprioceptive neuromuscular fasilition techniques (Other): No exercise intervention was made.
  Interventions: Other: Exercise, proprioceptive neuromuscular fasilition (PNF) techniques

INTERVENTIONS:
Other: Exercise, proprioceptive neuromuscular fasilition (PNF) techniques — PNF applications are defined as the autogenous inhibition, reciprocal inhibition, stress relaxation and gate control theory. Anterior elevation / posterior depression will be performed in the form of repetitive contractions using anterior depression / posterior elevation patterns. There will be 10 repetitions, with a 2-minute rest break between each technique. The treatment will continue twice a week for a total of 6 weeks.

SUMMARY:
Scapular dyskinesis is defined as the loss of strength around the scapular muscle, tightness of the pectoralis minor and disruption of scapular movements. Scapular patterns of proprioceptive neuromuscular fasilition (PNF) techniques are often preferred in the rehabilitation of scapular dyskinesis. The main principals of PNF applications are defined as the autogenous inhibition, reciprocal inhibition, stress relaxation and gate control theory.The aim of this study was to investigate the effect of scapular PNF patterns on muscular strength and pectoralis minor tightness among individuals with unilateral scapular dyskinesis.

DETAILED DESCRIPTION:
In order to standardize the measurements while evaluating individuals, the evaluation order will be as follows; The evaluation of minor pectoralis shortness, scapular dyskinesia by video analysis, scapular side shift test and then muscle strength evaluation will be done. The evaluation will be repeated before and 6 weeks after treatment and 12 weeks after treatment.

Proprioceptive Neuromuscular Facilitation Application:

Anterior elevation / posterior depression will be performed in the form of repetitive contractions using anterior depression / posterior elevation patterns. There will be 10 repetitions, with a 2-minute rest break between each technique. The treatment will be continued twice a week for a total of 6 weeks. Perceived Effort Scale, which is graded between 0-10, will be used to determine the level of perceived resistance to individuals before each treatment. In order to ensure standardization, the perceived effort level will be set to 5-6 (moderate).

ELIGIBILITY:
Inclusion Criteria:

* To be in the age range of 18-30,
* Being a sedentary,
* Having type 1 or type 2 scapular dyskinesia.

Exclusion Criteria:

* Has shoulder pain,
* Acute orthopedic injuries in the last 3 weeks, involving the upper extremity,
* Having had upper extremity surgery.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Upper trapez and serratus anterior muscle strength ratio and upper trapez and lower trapez muscle strength ratio | 12 weeks
  UT and SA muscle strength ratio (UT/SA) and UT and LT muscle strength ratio (UT/LT) were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Guney Deniz, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Other, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balci NC, Yuruk ZO, Zeybek A, Gulsen M, Tekindal MA. Acute effect of scapular proprioceptive neuromuscular facilitation (PNF) techniques and classic exercises in adhesive capsulitis: a randomized controlled trial. J Phys Ther Sci. 2016 Apr;28(4):1219-27. doi: 10.1589/jpts.28.1219. Epub 2016 Apr 28. PMID 27190456